CLINICAL TRIAL: NCT04653181
Title: Preoperative i.v. Iron Substitution in Patients With Colon Carcinoma and Iron-deficiency Anemia
Brief Title: Preoperative i.v. Iron Substitution in Patients With Colon Cancer
Acronym: PREFECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Selja Koskensalo, Consultant, abdominal surgeon,Md, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKoskensalo
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer
Keywords: postoperative complications
MeSH Terms: conditions — Colonic Neoplasms; Postoperative Complications | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron arm (Experimental): Half of patients get i.v. iron preoperatively
  Interventions: Drug: Ferric carboxymaltose
- non-iron arm (No Intervention): Half of patients are treated without i.v. iron substitution

INTERVENTIONS:
Drug: Ferric carboxymaltose — Iron-arm treated with Ferric carboxymaltose, non-iron arm without
  Other Names: Ferinject (intravenous iron )
  Arms: Iron arm

SUMMARY:
About 70% of colon cancer patients are anemic. Preoperative anemia in patients with colorectal cancer is associated with both impaired disease-free survival and overall survival. The purpose of this study is to compare the effects of preoperative iv iron substitution on postoperative recovery in preoperatively anemic (male Hb <130, female Hb <120) and iron deficient colon cancer patients in a prospective setup. As a primary outcome, the effect of iv-iron substitution on postoperative complications is investigated.

DETAILED DESCRIPTION:
Randomized preoperative iron substitution for patient with iron deficient anemia

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Dg: Colon ca
* The planned measure: the colon resection
* Men: Hb <130, women: Hb <120 and iron deficiency (elevated TfR, low TrFesat or low ferritin)

Exclusion Criteria:

* hyperreactivity for Ferinject
* haemochromatosis
* refusal for participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 30 days
  At study, difference between arms will be evaluated: Complications are analysed using Clavien-Dindo classification https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1360123/bin/3TT1.jpg

SECONDARY OUTCOMES:
Need for red blood cell transfusion | 30 days
  Number of Participants in need for red blood cells transfusion per arm

CONTACTS AND LOCATIONS:
Overall Officials: Selja K Koskensalo, Md, PhD, Study Director — Abdominal centre, HUCH
Locations (1):
- Jorvi Hospital, Espoo, HUS, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhen L, Zhe S, Zhenning W, Zhifeng M, Zhidong L, Xiaoxia L, Jianguang Y, Huimian X. Iron-deficiency anemia: a predictor of diminished disease-free survival of T3N0M0 stage colon cancer. J Surg Oncol. 2012 Mar 15;105(4):371-5. doi: 10.1002/jso.22032. Epub 2011 Jul 14. PMID 21761412
- [Background] Calvet X, Gene E, AngelRuiz M, Figuerola A, Villoria A, Cucala M, Mearin F, Delgado S, Calleja JL. Cost-minimization analysis favours intravenous ferric carboxymaltose over ferric sucrose or oral iron as preoperative treatment in patients with colon cancer and iron deficiency anaemia. Technol Health Care. 2016;24(1):111-20. doi: 10.3233/THC-151074. PMID 26409561
- [Background] Calleja JL, Delgado S, del Val A, Hervas A, Larraona JL, Teran A, Cucala M, Mearin F; Colon Cancer Study Group. Ferric carboxymaltose reduces transfusions and hospital stay in patients with colon cancer and anemia. Int J Colorectal Dis. 2016 Mar;31(3):543-51. doi: 10.1007/s00384-015-2461-x. Epub 2015 Dec 22. PMID 26694926
- [Background] Ristescu I, Pintilie G, Filip D, Jitca M, Fecheta R, Florescu I, Scripcariu V, Filipescu D, Grigoras I. Perioperative Anemia and Transfusion in Colorectal Cancer Patients. Chirurgia (Bucur). 2019 Mar-Apr;114(2):234-242. doi: 10.21614/chirurgia.114.2.234. PMID 31060656
- [Background] Dunne JR, Gannon CJ, Osborn TM, Taylor MD, Malone DL, Napolitano LM. Preoperative anemia in colon cancer: assessment of risk factors. Am Surg. 2002 Jun;68(6):582-7. PMID 12079143
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542